CLINICAL TRIAL: NCT03286725
Title: Physical Exercise for Education ('Fit to Study')
Acronym: FTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Helen Dawes, Principal Investigator, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EEF2681
Record Dates: First submitted 2017-08-16; First posted 2017-09-18 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Physical Activity; Mental Health Wellness 1; Cognitive Function 1, Social; Academic Attainment; Fitness Testing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: Single blind (outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The Control Group will be asked to continue with their normal PE lessons.
- Intervention Group (Experimental): 'Physical Education (PE) Programme'
  Interventions: Behavioral: Physical Education (PE) Programme

INTERVENTIONS:
Behavioral: Physical Education (PE) Programme — A programme of activities for PE lessons has been developed by Oxford Brookes University (in collaboration with Oxfordshire Sport and Physical Activity) to try to optimise the benefit of PE for brain function. Staff from Oxford Brookes University will train PE teachers to deliver this programme.
  The Intervention involves roughly 20 minutes of prescribed activities per week, to be delivered within school PE lessons.
  Arms: Intervention Group

SUMMARY:
Neuroscience evidence suggests that physical exercise can influence brain function and structure, both immediately and in the long-term. The 'Fit to Study' project is a randomised controlled trial to test the effects on academic performance (as well as fitness, wellbeing and cognitive function) of a teacher-training intervention designed to optimise the content of PE for brain and cognitive function during secondary school (Year 8) Physical Education (PE) lessons. The project aims to rigorously test the impact of this intervention in 100 state-funded secondary schools.

DETAILED DESCRIPTION:
Physical exercise has been shown to have positive effects on the brain and to improve cognitive performance, both immediately and in the long-term. This project is being conducted to understand better how the content of school PE, focusing on Year8 pupils during the academic year 2017/18, affects brain function and structure, and academic performance.

A programme of activities for PE lessons has been developed by Oxford Brookes University (in collaboration with Oxfordshire Sport and Physical Activity) to try to optimise the benefit of PE for brain function. Staff from Oxford Brookes University will train PE teachers to deliver this programme.

'Fit to Study' is aiming to recruit 100 state-funded secondary schools from within a radius of Oxford.

The National Foundation for Education Research will help with recruitment by sending materials to target schools, collating responses, collecting pupil information from schools that sign up, and passing information to the research teams and NatCen Social Research (who will be responsible for randomisation). Participating schools will be randomly assigned to either an Intervention Group (IG) and be asked to deliver the new PE programme, or to a Control Group (CG) and asked to continue with their normal PE lessons. Randomisation will be achieved using a random sequence generated using Stata12. Balance between treatment and control groups will be achieved across a range of covariates (i.e. to ensure not all girls schools are assigned to one condition).

For both Groups there will be a number of activities for schools to undertake, both at the start, during, and at the end of the study. The key tasks are listed, and then described, below:

* Online Cognitive Tests (pre- and post-study)
* Wellbeing Questionnaires (pre- and post-study)
* Physical Activity Assessments (before and during the study)
* PE Teacher Training for Intervention Schools
* Fitness (Beep) Tests (pre- and post-study)
* NatCen will undertake an Independent Evaluation of the 'Fit to Study' programme.

In all schools, the pupils in the target year group will undergo baseline assessments (in the final term of Year 7), which will comprise tests of physical fitness; cognitive assessments; and questionnaires (about physical activity, sleep patterns, mood, motivation and wellbeing). The tests of physical fitness will be administered during PE lessons and will involve measures of speed and endurance. The school PE teachers will be involved in the administration of these tests. The cognitive tests (which will include tests of memory, executive functions and attention using button responses), and some of the questionnaires, will be computer-based and may be administered over the web, at school or at home, using a well-established online testing package.

PE teachers in the intervention condition schools will be trained to administer our intervention. Our training package will comprise a set of focused lesson principles and techniques for their delivery.

To foster friendly competition between schools, the investigators may produce newsletters/bulletins containing school league tables indicating summary physical activity levels during PE and/or proportion of assessments completed, but these will never contain individual pupils' data.

The investigators will use activity monitors to compare physical activity during intervention and control PE lessons. At the end of the intervention period (which is intended to be an academic year), the Year 8 pupils in all schools will repeat the assessments.

In addition, the University of Oxford will be conducting a sub-study with a small number of pupils from a subset of schools. This is an optional part of the project and will be subject to separate written / informed consent from the pupils' parents/guardians. This will involve MRI brain scanning at the University of Oxford, as well as additional fitness and cognitive tests. Further detail will be made available to schools that are selected to take part in the Main Study (from May 2017).

ELIGIBILITY:
Inclusion Criteria:

Inclusion is by school year group - typically aged 11-14:

* Year 7 pupils during the academic year 2016/17 (Age 11-12, KS3).
* Year 8 pupils during the academic year 2017/18 (Age 12-13, KS3).

Exclusion Criteria:

* Any pupils that are exempted from PE.
* Pupils that have 'opted out' of data sharing / storage for research purposes

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Mathematical attainment: as measured using the level 13 Progress in Maths test (provided at GL assessment) at the end of the school year (June 2018). | 1 hour: Last month of the study (June 2018).
  The Primary Outcome Measure is recorded on the ISRCTN registry with study ID ISRCTN15730512.
  Mathematical attainment as measured using the level 13 Progress in Maths test (provided at GL assessment) at the end of the school year.

SECONDARY OUTCOMES:
Wellbeing Survey | 30 minutes: Baseline (June 2017) and final month of the study (June 2018)
  A battery of surveys each including a number of measures: adolescent mental health and wellbeing; daytime sleepiness; physical and global self-esteem; PE enjoyment; single measures of health-related quality of life and weekly moderate to vigorous physical activity (MVPA); attitudes, social norms, competence, intentions and willingness in relation to physical activity. Approximately 60 questions in total, taking 30 minutes to complete.
Cognitive Test of Attention and Reaction Time | 10 minutes: Baseline (June 2017) and final month of the study (June 2018)
  This is one of five (computer-based) cognitive tasks developed via jsPsych that are completed by participants at one sitting. It is an attention/ reaction-time task, to appearance of red triangles on the screen.
Cognitive Test of Memory (Image Associates) | 10 minutes: Baseline (June 2017) and final month of the study (June 2018)
  This is one of five (computer-based) cognitive tasks developed via jsPsych that are completed by participants at one sitting. It is an (image) association of place, person and object (memory) task.
Eriksen Flanker Test | 10 minutes: Baseline (June 2017) and final month of the study (June 2018)
  This is one of five (computer-based) cognitive tasks developed via jsPsych that are completed by participants at one sitting. It is a (modified) Eriksen Flanker task.
Cognitive Test of Memory (Two-back Image Task) | 10 minutes: Baseline (June 2017) and final month of the study (June 2018)
  This is one of five (computer-based) cognitive tasks developed via jsPsych that are completed by participants at one sitting. It is a two-back image (memory) task (saying whether a picture is the same as the one before last).
Cognitive Test of Executive Function | 10 minutes: Baseline (June 2017) and final month of the study (June 2018)
  This is one of five (computer-based) cognitive tasks developed via jsPsych that are completed by participants at one sitting. It is a task-switching (executive function) task (arms up or arms down characters in relation to shape or colour questions).
Fitness Assessment (20m Beep Test) | 20 minutes: Baseline (June 2017) and final month of the study (June 2018)
  A distance of 20m is measured; cones are placed at lines indicating the distance. Pupils stand behind one of the lines facing the 2nd line, and begin running when instructed by an audio recording. The pupils continue running between the two lines, turning when signalled by the recorded beeps. After one minute, a sound indicates an increase in speed, and the beeps will be closer together. This continues each minute (level). If the line is reached before the beep sounds, the subject must wait until the beep sounds before continuing. If the line is not reached before the beep sounds, the subject is given a warning and must continue to run to the line, then turn and try to catch up with the pace within two more 'beeps'. The test is stopped if the subject fails to reach the line (within 2m) for two consecutive ends after a warning. Participants are instructed to remember the last number that was called before they stopped and tell the teacher who is recording the scores.
Physical Activity Measurements | 60 minutes: Baseline (June 2017), at 14 weeks, at 28 weeks and final month of the study (June 2018).
  All pupils will be provided with wrist-worn Axivity AX3 accelerometers, to be worn on the non-dominant wrist, to record their physical activity (PA) during a PE lesson. The AX3 is a tri-axial accelerometer which measures linear acceleration from +/- 2g to +/- 16g range along three orthogonal axes known as 'z' (upward and downward), 'y' (left and right) and 'x' (forward and backward).

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
On conclusion of the project, the Fischer Family Trust (see http://www.fft.org.uk/) will collate and upload anonymised data to the UK Data Archive (for the primary outcome measure). This archived data (for the primary outcome measure) will only be available in an anonymised form with restricted access for research purposes only.

REFERENCES:
- [Derived] Wassenaar TM, Wheatley CM, Beale N, Nichols T, Salvan P, Meaney A, Atherton K, Diaz-Ordaz K, Dawes H, Johansen-Berg H. The effect of a one-year vigorous physical activity intervention on fitness, cognitive performance and mental health in young adolescents: the Fit to Study cluster randomised controlled trial. Int J Behav Nutr Phys Act. 2021 Mar 31;18(1):47. doi: 10.1186/s12966-021-01113-y. PMID 33789683
- [Derived] Beale N, Eldridge E, Delextrat A, Esser P, Bushnell O, Curtis E, Wassenaar T, Wheatley C, Johansen-Berg H, Dawes H. Exploring activity levels in physical education lessons in the UK: a cross-sectional examination of activity types and fitness levels. BMJ Open Sport Exerc Med. 2021 Mar 9;7(1):e000924. doi: 10.1136/bmjsem-2020-000924. eCollection 2021. PMID 33768961
- [Derived] Wassenaar TM, Wheatley CM, Beale N, Salvan P, Meaney A, Possee JB, Atherton KE, Duda JL, Dawes H, Johansen-Berg H. Effects of a programme of vigorous physical activity during secondary school physical education on academic performance, fitness, cognition, mental health and the brain of adolescents (Fit to Study): study protocol for a cluster-randomised trial. Trials. 2019 Apr 2;20(1):189. doi: 10.1186/s13063-019-3279-6. PMID 30940164